CLINICAL TRIAL: NCT05656521
Title: A Prospective, Randomized, Comparative, Multi-centric, Adaptive Design Clinical Study to Evaluate Efficacy, Safety, and Tolerability of 101-PGC-005 ('005) for the Treatment of Moderate Corona Virus Disease (COVID-19) Patients
Brief Title: 101-PGC-005 for the Treatment of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: 101 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PGC-005-IN-101-2
Record Dates: First submitted 2022-12-13; First posted 2022-12-19 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19; Infectious Disease; Dexamethasone; Inflammation; Cytokine Storm
MeSH Terms: conditions — COVID-19; Communicable Diseases; Inflammation; Cytokine Release Syndrome | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- '005 Treatment Arm (Experimental): '005 IV 20 mg + Standard of care
  Interventions: Drug: 101-PGC-005
- Dexamethasone Treatment Arm (Active Comparator): Dexamethasone 6 mg + Standard of care
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: 101-PGC-005 — '005 is a targeted prodrug of dexamethasone that binds to activated macrophages.
  Arms: '005 Treatment Arm
Drug: Dexamethasone — Dexamethasone is a glucocorticoid commonly prescribed to treat inflammation.
  Arms: Dexamethasone Treatment Arm

SUMMARY:
This is a prospective, randomized, comparative, multi-centric, adaptive design clinical study to evaluate efficacy, safety, and tolerability of 101-PGC-005 ('005) when used alongside standard of care (SOC) for the treatment of hospitalized patients with coronavirus disease (COVID-19).

DETAILED DESCRIPTION:
The study is planned as an adaptive Phase II/III clinical study to allow for seamless transition to Phase III after completion of Phase II. The study will begin as initially only a Phase II to evaluate and compare the efficacy, safety, and tolerability of bolus injection of 20 mg '005 vs dexamethasone 6 mg injection for the treatment of COVID-19.

The treatment period with the investigational product in the test group will be 3 consecutive days. However, in the comparator group, the patient will be allowed to take 6 mg dexamethasone daily for the duration of their treatment, based on the investigator's clinical judgement for a total of not more than 10 days or until the time of discharge, whichever is earlier. All patients in either test or control groups will be allowed to take other concomitant SOC as per the prescribed schedule for entire duration of the study, as applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of age 18 to 65 years (both inclusive) who have been hospitalized for treatment of moderate COVID-19 disease.
2. Patients with 'moderate' COVID-19 disease severity, as defined by Comprehensive Guidelines for Management of COVID-19 patients, Directorate General of Health Services, MoHFW, GOI; AND having any of the following symptoms and signs prior to randomization:

   1. Fever, cough, with or without sore throat/throat irritation, body ache/headache, malaise/weakness, diarrhoea or gastrointestinal upset, with or without anorexia/nausea/vomiting, with or without loss of smell and/or taste, shortness of breath/breathlessness and difficulty in breathing
   2. Respiratory rate of >24 to <30 breaths/min,
   3. SpO2: 90 - 93% on room air
3. Patients with positive RT-PCR test for SARS-CoV-2 in nasopharyngeal or oropharyngeal swabs (sample collected within 7 days prior to randomization)
4. Elevated CRP, ESR or Ferritin levels
5. In case of female patients of child-bearing potential, a negative urine pregnancy test prior to beginning the therapy.
6. Willing to sign voluntary informed consent for participation in the study and willing to adhere to all protocol procedures. In case the subject is unable to provide informed consent than the same should be obtained from legally acceptable representative (LAR).

Exclusion Criteria:

1. Patients with 'mild' or 'severe' COVID-19 disease severity, as defined by latest Comprehensive Guidelines for Management of COVID-19 patients, Directorate General of Health Services, MoHFW, GOI at the time of randomization. This includes any one or more of the following

   1. Peripheral Blood oxygen saturation ≥94% or <90%
   2. Respiratory Rate or <24 or ≥30 breaths per minute
2. First positive RT-PCR more than 7 days prior to treatment administration
3. Patients with evidence of other serious infectious, malignant, autoimmune, kidney, hepatic, cardiovascular or other systemic disease and/or laboratory abnormality, which, in the opinion of the investigator, prevent the patient from participating in the study
4. Subjects with Chronic liver disease (Child Pugh class B or C) and chronic renal disease (GFR<30ml/min).
5. Renal dysfunction [Serum Creatinine > 2.5 times of ULN or calculated creatinine clearance < 30ml/min], Liver Dysfunction [Total Bilirubin > 3times ULN & AST/ALT > 5times ULN].
6. Chronic systemic glucocorticoid treatment or any immunosuppressive treatment
7. History of human immunodeficiency virus (HIV) or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
8. Pregnant and Lactating patients.
9. Patients who require IL-6 inhibitors for management of inflammation at the time of study entry.
10. Subject has a psychiatric disease that is not well controlled where controlled is defined as: stable on a regimen for more than one year.
11. Hospital discharge is anticipated in ≤ 24 hours or anticipated transfer to another hospital which is not a study site within 72 hours.
12. Patients that are currently or have participated in such studies participating in other clinical studies with investigational drug, biological agent or device within 1 month or within 5 half-lives (of the drug/biologic) prior to randomization (whichever is longer).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement | Baseline through Days 10, 14, 28
  Clinical improvement or shift in WHO 11-point ordinal scale rating

SECONDARY OUTCOMES:
Reduction in Symptoms | Baseline through Days 10, 14, 28
  Improvement in COVID-19 Symptoms such as fever, heart rate, and oxygen saturation
Reduction in Inflammatory Markers | Baseline and Days 14, 28
  Improvement in biochemical inflammatory markers such as CRP, Neutrophil-Lymphocyte (N/L) ratio, D-Dimer, Sr. Ferritin, IL-6, and TNF-α
Reduction in Oxygen Supplementation | 28 days
Discharge Rate from hospital | 28 days
Reduction in ICU Admission/Mechanical Ventilation | 28 days
Reduction in time to Respiratory Viral Clearance | Days 3, 7, 10, 14
Reduction in Lung Injury on Chest HRCT | Baseline and 14, 28 Days
Reduction in All-cause Mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Government Medical College & General Hospital, Srikakulam, Andhra Pradesh
  - Victoria Hospital Bangalore, Bangalore, Karnataka
  - Sangvi Multispeciality Hospital, Pune, Maharashtra
  - SMS Medical College and Attached Hospitals, Jaipur, Rajasthan
  - Santosh Medical College and Hospital, Ghaziabad, Uttar Pradesh